CLINICAL TRIAL: NCT01260285
Title: The Safety of Vardenafil in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: McGuire Research Institute (Other)
Responsible Party: Dr. Ion Jovin, MD, McGuire VAMC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01703
Record Dates: First submitted 2010-12-10; First posted 2010-12-15 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-11

CONDITIONS: Ischemia-reperfusion Injury.
MeSH Terms: conditions — Reperfusion Injury | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vardenafil (Experimental)
  Interventions: Drug: Vardenafil

INTERVENTIONS:
Drug: Vardenafil — 10 mg PO once

SUMMARY:
The purpose of this study is to evaluate the safety of vardenafil in cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* undergoing cardiac surgery

Exclusion Criteria:

* emergent surgery
* recent MI in past 7 days prior to surgery
* ejection fraction < 35%
* creatinine > 2.0
* prior CVA
* severe COPD
* recent use of nitrates (within past 48 hours prior to surgery)
* prior CABG
* pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Hypotension | approximately 5 days

SECONDARY OUTCOMES:
Ejection Fraction | approximately 5-7 days postop

CONTACTS AND LOCATIONS:
Overall Officials: Ion Jovin, MD, Principal Investigator — McGuire VAMC
Locations (1):
- McGuire VAMC, Richmond, Virginia, United States